CLINICAL TRIAL: NCT04001166
Title: Pharmacogenomics of Antithrombotic Drugs (PreMed PGx Study)
Brief Title: Pharmacogenomics of Antithrombotic Drugs -a Register Linkage Study With National Registries and Biobanks in Finland
Status: Completed | Type: Observational
Sponsor: VTT Technical Research Centre of Finland (Other)
Collaborators: Helsinki Biobank (Unknown); THL Biobank (Unknown); Auria Biobank (Unknown); Hospital District of Helsinki and Uusimaa (Other); Hospital District of Southwestern Finland (Other); Finnish Institute for Health and Welfare (Other Government); Social Insurance Institution, Finland (Other)
Responsible Party: Sponsor
Other Study IDs: PreMed
Record Dates: First submitted 2019-05-28; First posted 2019-06-27 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Individuals With a Disease of Cardiovascular System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Non-interventional study — This is a non-interventional study. Patients will be treated with any treatment deemed appropriate by the patient's physician.

SUMMARY:
This is a retrospective cohort study linking data from Finnish Biobanks (Helsinki Biobank, Auria Biobank and THL Biobank), laboratory databases, and national registries of Social Insurance Institution of Finland (Kela) and the National Institute of Health and Welfare (THL) to investigate pharmacogenomics of antithrombotic drugs in the Finnish population. The purpose of the study is to assess clinical and economic aspects of using genomic data in the context of antithrombotic drug therapy.

Based on earlier research, data regarding variant alleles in CYP2C9 and VKORC1 will be used in the primary analyses. Individuals with and without specific variant alleles are compared in respect to their clinical response to warfarin therapy. Warfarin-treated individuals are also analysed in relation to other clinical outcomes and a wide range of healthcare encounters.

The explorative part of the study will employ data-driven classification methods to explore genotype-phenotype associations for a larger group of antithrombotic drugs including direct oral anticoagulants, clopidogrel and heparins and possible interactions with other drugs. In this part, 26 gene variants identified in literature will be used.

The retrospective follow-up time for the study participants is from January 2007 to December 2018, or 2 years prior the first anticoagulant drug is purchased until 6 months after the last purchase.

ELIGIBILITY:
Inclusion Criteria:

* Genotyped for CYP2C9/rs1799853, CYP2C9/rs1057910 and VKORC1/rs9923231
* Diagnosed with at least one of the following:

  * Atrial Fibrillation and Flutter (I48)
  * Ischemic Heart Disease (I20-I25)
  * Cerebrovascular disease (I63,I65,I66, 167.2, I69.3-I69.8)
  * Atherosclerosis (I70)
  * Pulmonary embolism (I26)
  * Phlebitis and thrombophlebitis (I80)
  * Portal vein thrombosis (I81)
  * Other venous embolism and thrombosis (I82)
* Purchased at least one of the following drugs between January 1st 2007 - December 31st 2018:

  * Anticoagulants: Warfarin, Dabigatran, Apixaban, Rivaroxaban, Edoxaban, Heparin, Enoxaparin, Dalteparin
  * Antiplatelets: Clopidogrel, Ticagrelor, Acetylsalicylic acid

Exclusion Criteria:

* Permanent residence in Finland less than 12 months during the follow-up period
* Purchase of any of the antithrombotic drugs listed above between January 1st 2005 - December 31st 2006

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of adults diagnosed with a disease of cardiovascular system and genotyped for variants in CYP2C9 and VKORC1, and who have used antithrombotic drugs between January 1st 2007 - December 31st 2018.
Sampling Method: Non-Probability Sample
Enrollment: 7005 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2020-04-28 (Actual); Study Completion 2020-04-28 (Actual)

PRIMARY OUTCOMES:
Incidence of bleeding complications | During warfarin treatment and beyond 6 months after the treatment
  Incidence of bleeding complications in warfarin-treated individuals

SECONDARY OUTCOMES:
Time in Therapeutic Range (TTR) | During warfarin treatment and beyond 6 months after the treatment
  TTR during first three months in warfarin-treated individuals
Time to reach therapeutic range | During warfarin treatment and beyond 6 months after the treatment
  Time to reach therapeutic range in warfarin-treated individuals
Time-weighted mean INR | During warfarin treatment and beyond 6 months after the treatment
  INR (time-weighed mean) during the first month in warfarin-treated individuals
Incidence of outpatients visits | During warfarin treatment and beyond 6 months after the treatment
  Incidence of outpatient visits caused by bleeding in warfarin-treated individuals
Incidence of laboratory visits | During warfarin treatment and beyond 6 months after the treatment
  Incidence of laboratory visits related to warfarin treatment in warfarin-treated individuals
The number of laboratory tests | During warfarin treatment and beyond 6 months after the treatment
  The number of performed laboratory tests laboratory tests related to warfarin treatment in warfarin-treated individuals
Incidence of emergency room (ER) visits | During warfarin treatment and beyond 6 months after the treatment
  Incidence of ER visits caused by bleeding, myocardial infarction or cerebral infarction in warfarin-treated individuals
Indicidence of hospital admissions | During warfarin treatment and beyond 6 months after the treatment
  Hospitalizations caused by bleeding, myocardial infarction or cerebral infarction in warfarin-treated individuals
The number of hospital inpatient days | During warfarin treatment and beyond 6 months after the treatment
  The number of inpatient days caused by bleeding, myocardial infarction or cerebral infarction in warfarin-treated individuals
Incidence of medical procedures | During warfarin treatment and beyond 6 months after the treatment
  Incidence of medical procedures caused by bleeding, myocardial infarction or cerebral infarction in warfarin-treated individuals

CONTACTS AND LOCATIONS:
Overall Officials: Jari Ahola, Study Director — VTT Technical Research Centre of Finland; Mark van Gils, PhD, Principal Investigator — VTT Technical Research Centre of Finland
Locations (1):
- To learn more about this study, you or your doctor may contact the study research staff using the contact information provided by the sponsor., Multiple Locations, Finland

REFERENCES:
- [Derived] Vuorinen AL, Lehto M, Niemi M, Harno K, Pajula J, van Gils M, Lahteenmaki J. Pharmacogenetics of Anticoagulation and Clinical Events in Warfarin-Treated Patients: A Register-Based Cohort Study with Biobank Data and National Health Registries in Finland. Clin Epidemiol. 2021 Mar 8;13:183-195. doi: 10.2147/CLEP.S289031. eCollection 2021. PMID 33727862
- See also: Related Info — http://www.vtt.fi/premed